CLINICAL TRIAL: NCT06903442
Title: Developing a Brief Intervention to Communicate Cardiovascular Risk to Patients Presenting to the Emergency Department With Chest Pain: a Co-Production Approach. Phase 2.
Acronym: ACTION 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AC25029
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients assigned to usual clinical care
- Intervention (Experimental): Patients will return to outpatients department to receive a cardiovascular brief intervention
  Interventions: Behavioral: Co-designed cardiovascular brief intervention

INTERVENTIONS:
Behavioral: Co-designed cardiovascular brief intervention — Patients will be randomised to a brief intervention where they will be informed of their high-sensitivity cardiac troponin value and cardiovascular risk.
  Arms: Intervention

SUMMARY:
Some patients who come to the emergency department with chest pain and have not had a heart attack, are at an increased risk of having a heart attack in the future. The investigators know this by taking a blood test (troponin) which looks at damage to the patient's heart.

These patients are often sent home from hospital with no information about their risk of heart disease. A patient survey revealed that patients in the emergency department would like to receive more information about heart disease.

In this study the investigators will provide patients who are at increased risk of cardiovascular disease with their troponin value. The investigators will deliver this information within a cardiovascular brief intervention, which is a short conversation with a patient about their health. In a previous study the investigators carried out some interviews with patients to find out how their results should be delivered and what information should be included in a cardiovascular brief intervention. The investigators also asked them the best way to provide patients with this information. The aim of this part of the study it to determine if the new cardiovascular brief intervention helps patients understand their risk and if it results in them making changes to their health.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the Emergency Department with symptoms suggestive of acute coronary syndrome
* A maximum high-sensitivity cardiac troponin I between 5 ng/L and the sex-specific 99th centile.
* Resides in Scotland and has a CHI number
* Adults aged 18 and over
* No history of cardiovascular disease
* At least 1 modifiable cardiovascular risk factor: current smoker, hypertension (140/90 mmHg), hypercholesterolaemia (>6.0 mmol/L), overweight and obesity (BMI >25), hyperglycaemia or diabetes mellitus.
* Patients who are able to provide informed consent

Exclusion Criteria:

* Patients with a diagnosis of acute coronary syndrome during index presentation
* Patients who are not able to give informed consent
* Patients who do not speak English
* Patients who are unable to attend hospital as outpatient to receive the cardiovascular brief intervention
* Patients with ongoing or planned cardiovascular investigations or interventions
* Patients with chronic kidney disease and a eGFR below 30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Health | 90 days
  Cardiovascular health will be measured using a lifestyle questionnaire based on the American Heart Association's Life's Essential 8 measure of cardiovascular health (Lloyd-Jones, 2022). The components of Life's Essential 8 include (diet, physical activity, nicotine exposure, body mass index, sleep, blood pressure, blood glucose and blood cholesterol). Each component has a scoring metric of 0-100 (table 1) with a composite score of cardiovascular health being the average of all 8 components. A higher score represents better cardiovascular health.

SECONDARY OUTCOMES:
High sensitivity cardiac troponin concentrations | 90 days
  High-sensitivity cardiac troponin I will be assessed as an absolute value and change between baselines and 90 days for the secondary objective. Additional exploratory analyses will evaluate other high-sensitivity cardiac troponin assays and measures.
Motivational readiness to make changes to improve their cardiovascular health | 90 days
  Patient's motivation will be assessed using a "readiness ruler" linear numeric scale (0-10)
The difference in scores within each component of the Life's Essential 8 cardiovascular health score | 90 days
  Cardiovascular health will be measured using a lifestyle questionnaire based on the American Heart Association's Life's Essential 8 measure of cardiovascular health (Lloyd-Jones, 2022). The components of Life's Essential 8 include (diet, physical activity, nicotine exposure, body mass index, sleep, blood pressure, blood glucose and blood cholesterol).

OTHER OUTCOMES:
Cardiac medication adherence | 90 days
  Medication use and adherence will be assessed using the Medication Adherence Reporting Scale (MARS-5) (Horne 1999). The participants will rate 5 different adherence behaviours on a five-point scale. The scores are combined to provide a total score, with the higher scores indicating a higher level of reported adherence to medication.
Proportion of participants recruited from screening log | 90 days
  Recruitment rates and patients lost to follow up will be assessed from the trial consort diagram which will detail the participants' pathway though the study.
The quantity of missing data at baseline and follow up | 90 days
  The proportion of missing data will be assessed from the case report forms.
The presence or increase of anxiety and/or depression | 90 days
  Anxiety and depression will be assessed using the Hospital and Anxiety Depression Scale (HADS) (Zigmond and Snaith 1983). The HADS consists of 14 questions which can be scored from 0 to 3. Anxiety and depression are scored separately with a maximum score of 21 for each category.
Patient's acceptability and views of the cardiovascular brief intervention | 120 days
  will be explored through qualitative interviews with patients

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the primary paper, a deidentified individual participant data set will be will be made available for data sharing purposes, subject to necessary governance approvals. Access to the deidentified dataset will be under a controlled access model.
Supporting Information: Study Protocol, ICF